CLINICAL TRIAL: NCT02057133
Title: A Phase 1b Study of Abemaciclib in Combination With Therapies for Patients With Metastatic Breast Cancer
Brief Title: A Study of LY2835219 (Abemaciclib) in Combination With Therapies for Breast Cancer That Has Spread
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15252; I3Y-MC-JPBH (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Letrozole; Anastrozole; Tamoxifen; exemestane; Everolimus; Trastuzumab; LY3023414; Fulvestrant; pertuzumab; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- LY2835219 + Letrozole (Experimental): LY2835219 administered orally. Letrozole administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Letrozole
- LY2835219 + Anastrozole (Experimental): LY2835219 administered orally. Anastrozole administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Anastrozole
- LY2835219 + Tamoxifen (Experimental): LY2835219 administered orally. Tamoxifen administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Tamoxifen
- LY2835219 + Exemestane (Experimental): LY2835219 administered orally. Exemestane administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Exemestane
- LY2835219 + Exemestane + Everolimus Dose Escalation (Experimental): LY2835219 administered orally. Exemestane administered orally. Everolimus administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Exemestane; Drug: Everolimus
- LY2835219 + Exemestane + Everolimus Dose Expansion (Experimental): LY2835219 administered orally. Exemestane administered orally. Everolimus administered orally. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Exemestane; Drug: Everolimus
- LY2835219+ Trastuzumab Dose Escalation (Experimental): LY2835219 administered orally. Trastuzumab administered intravenously (IV) infusion. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Trastuzumab
- LY2835219+ Trastuzumab Dose Expansion (Experimental): LY2835219 administered orally. Trastuzumab administered IV infusion. This arm is closed to enrollment.
  Interventions: Drug: LY2835219; Drug: Trastuzumab
- LY3023414 + LY2835219 + Fulvestrant Dose Escalation (Experimental): LY3023414 administered orally. LY2835219 administered orally. Fulvestrant administered intramuscularly (IM).
  Interventions: Drug: LY2835219; Drug: LY3023414; Drug: Fulvestrant
- LY3023414 + LY2835219 + Fulvestrant Dose Expansion (Experimental): LY3023414 administered orally. LY2835219 administered orally. Fulvestrant administered IM.
  Interventions: Drug: LY2835219; Drug: LY3023414; Drug: Fulvestrant
- LY2835219 +Trastuzumab +Pertuzumab +Loperamide Dose Escalation (Experimental): LY2835219 administered orally. Loperamide administered orally. Trastuzumab administered IV infusion. Pertuzumab administered IV infusion.
  Interventions: Drug: LY2835219; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Loperamide
- LY2835219 +Trastuzumab + Pertuzumab +Loperamide Dose Expansion (Experimental): Hormone Receptor Negative (HR-): LY2835219 administered orally. Loperamide administered orally. Trastuzumab administered IV infusion. Pertuzumab administered IV infusion.
  Hormone Receptor Positive (HR+): LY2835219 administered orally. Loperamide administered orally. Trastuzumab administered IV infusion. Pertuzumab administered IV infusion. Endocrine therapy administered orally.
  Interventions: Drug: LY2835219; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Loperamide; Drug: Endocrine therapy
- LY2835219 + Endocrine Therapy (Experimental): LY2835219 administered orally. Ongoing endocrine therapy administered orally.
  Interventions: Drug: LY2835219; Drug: Endocrine therapy

INTERVENTIONS:
Drug: LY2835219 — Administered orally.
  Other Names: Abemaciclib
Drug: Letrozole — Administered orally.
  Arms: LY2835219 + Letrozole
Drug: Anastrozole — Administered orally.
  Arms: LY2835219 + Anastrozole
Drug: Tamoxifen — Administered orally.
  Arms: LY2835219 + Tamoxifen
Drug: Exemestane — Administered orally.
  Arms: LY2835219 + Exemestane; LY2835219 + Exemestane + Everolimus Dose Escalation; LY2835219 + Exemestane + Everolimus Dose Expansion
Drug: Everolimus — Administered orally.
  Arms: LY2835219 + Exemestane + Everolimus Dose Escalation; LY2835219 + Exemestane + Everolimus Dose Expansion
Drug: Trastuzumab — Administered IV infusion.
  Arms: LY2835219 +Trastuzumab + Pertuzumab +Loperamide Dose Expansion; LY2835219 +Trastuzumab +Pertuzumab +Loperamide Dose Escalation; LY2835219+ Trastuzumab Dose Escalation; LY2835219+ Trastuzumab Dose Expansion
Drug: LY3023414 — Administered orally.
  Arms: LY3023414 + LY2835219 + Fulvestrant Dose Escalation; LY3023414 + LY2835219 + Fulvestrant Dose Expansion
Drug: Fulvestrant — Administered IM.
  Arms: LY3023414 + LY2835219 + Fulvestrant Dose Escalation; LY3023414 + LY2835219 + Fulvestrant Dose Expansion
Drug: Pertuzumab — Administered IV infusion.
  Arms: LY2835219 +Trastuzumab + Pertuzumab +Loperamide Dose Expansion; LY2835219 +Trastuzumab +Pertuzumab +Loperamide Dose Escalation
Drug: Loperamide — Administered orally.
  Arms: LY2835219 +Trastuzumab + Pertuzumab +Loperamide Dose Expansion; LY2835219 +Trastuzumab +Pertuzumab +Loperamide Dose Escalation
Drug: Endocrine therapy — Endocrine therapy administered orally.
  Arms: LY2835219 + Endocrine Therapy; LY2835219 +Trastuzumab + Pertuzumab +Loperamide Dose Expansion

SUMMARY:
This study evaluates the safety of abemaciclib in combination therapies (letrozole, anastrozole, tamoxifen, exemestane, exemestane plus everolimus, trastuzumab, LY3023414 plus fulvestrant, pertuzumab plus trastuzumab with loperamide, or ongoing endocrine therapy) for breast cancer that has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of hormone receptor positive (HR+), human epidermal growth factor receptor 2 (HER2) negative metastatic breast cancer for Parts A to E, G, and I.
* Have a diagnosis of human epidermal growth factor receptor 2 (HER2) positive metastatic breast cancer for Parts F and H.
* For Part A (LY2835219 + letrozole): Except for ongoing therapy with letrozole, the participant must not have received prior systemic endocrine therapy for metastatic disease.
* For Part B (LY2835219 + anastrozole): Except for ongoing therapy with anastrozole, the participant must not have received prior systemic endocrine therapy for metastatic disease.
* For Part C (LY2835219 + tamoxifen): The participant may have received prior systemic endocrine therapy for metastatic disease and may be receiving ongoing therapy with tamoxifen.
* For Part D (LY2835219 + exemestane): The participant must have received prior systemic endocrine therapy with at least one nonsteroidal aromatase inhibitor (anastrozole, letrozole) for metastatic disease and may be receiving ongoing therapy with exemestane.
* For Part E (LY2835219 + exemestane + everolimus): The participant must have received prior systemic endocrine therapy with at least one nonsteroidal aromatase inhibitor (anastrozole, letrozole) for metastatic disease and may be receiving ongoing therapy with either exemestane or exemestane + everolimus.
* For Part F (LY2835219 + trastuzumab):The participant must have received at least 1 chemotherapy regimen for metastatic disease and may be receiving ongoing therapy with trastuzumab. The participant must have an estimated left ventricular ejection fraction within the normal range by either echocardiogram or multigated acquisition (MUGA) scan
* For Part G (abemaciclib + LY3023414 + fulvestrant): The participant may have received prior systemic endocrine therapy with at least one nonsteroidal aromatase inhibitor (anastrozole, letrozole) for metastatic disease.
* For Part H: (abemaciclib + trastuzumab + pertuzumab): The participant must have received at least 1 chemotherapy regimen for metastatic disease. The participant may be receiving ongoing therapy with trastuzumab and/or pertuzumab at the time of study entry. The participant must have an estimated left ventricular ejection fraction (LVEF) within the normal range by either echocardiogram or multigated acquisition (MUGA) scan.
* For Part I (abemaciclib + endocrine therapy): The participant must have demonstrated evidence of disease progression on a Cyclin Dependent Kinase 4 (CDK4) and Cyclin Dependent Kinase 6 (CDK6) inhibitor (either palbociclib or ribociclib) plus endocrine therapy for advanced or metastatic disease as the most recent therapy immediately preceding study entry. The participant should remain on the current endocrine therapy while receiving abemaciclib.
* For Parts A, B, C, D, E, and F: Have either measureable disease or nonmeasureable but evaluable bone disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* For Part G, H, and I: Have measureable disease as defined by RECIST 1.1.
* For all Parts except Part F and H: Participants must have either post-menopausal status or pre-menopausal status if continuing or beginning ovarian suppression with a luteinizing hormone-releasing hormone (LHRH) agonist such as goserelin.
* Parts H, and I: Must be able and willing to undergo mandatory tumor biopsies prior to study treatment and at the time of discontinuation from study treatment.
* Have adequate organ function, including:

  * Hematologic: Absolute neutrophil count (ANC) ≥1.5 x 10^9/liter (L), platelets ≥ 100 x 10^9/L, and hemoglobin ≥ 8 gram/deciliter (g/dL).
  * Hepatic: Bilirubin ≤1.5 times upper limits of normal (ULN), alanine aminotransferase (ALT) ≤ 3.0 times ULN.
  * Renal: Serum creatinine ≤ 1.5 times ULN.
* Have a performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for breast cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy), except for ongoing corresponding combination therapy, for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug(s), and recovered from the acute effects of therapy (until the toxicity resolves to either baseline or at least Grade 1) except for residual alopecia or peripheral neuropathy. For Part F and H: concurrent treatment with trastuzumab emtansine (T-DM1) is not allowed.

Exclusion Criteria:

* Have metastatic breast cancer with severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of the disease.
* Have brain metastasis without prior radiotherapy.
* For Parts A, B, C, D, E, G and I: Have received prior systemic chemotherapy for metastatic disease. However, the participant may have received prior systemic chemotherapy in the neoadjuvant or adjuvant setting.
* For Parts A, B, C, D, E, F, H: Have received prior therapy with a CDK4/6 inhibitor, Part G: Have received prior therapy with fulvestrant or any PI3K and/or mTOR inhibitor (including LY3023414); Part I: Have received prior treatment with abemaciclib in any setting.
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (including interstitial lung disease (ILD), severe dyspnea at rest or requiring oxygen therapy or, history of major surgical resection involving the stomach or small bowel).
* Have central nervous system (CNS) metastasis with either radiotherapy or development of neurological changes ≤14 days prior to receiving study treatment. Participants may be receiving a stable dose of corticosteroids. Screening of asymptomatic participants without history of CNS metastasis is not required. Untreated CNS metastases are not permitted.
* For Parts F and H: Cardiac disease including myocardial infarction within 6 months, unstable angina, or New York Heart Association (NYHA) Grade II or greater functional impairment.
* For Part G: Have type 1 diabetes mellitus or a history of gestational diabetes mellitus. Participants with a type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained with oral therapy as documented by Hemoglobin A1c <7%.
* For Part G: Have a baseline electrocardiogram (obtained from Day -14 to Day -1) with any of the following abnormal findings: ventricular arrhythmia, evidence of acute myocardial ischemia, heart block (of any degree), or QTc prolongation (defined as QTcB ≥450 milliseconds).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-03-10 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Drug-Related Adverse Events | Baseline through study completion (estimated as 12 months)
  Number of participants with one or more drug-related adverse events

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY2835219, Letrozole, Anastrozole, Tamoxifen, Exemestane, Everolimus, Trastuzumab, LY3023414, Fulvestrant, and Pertuzumab | Cycle 1 up to Cycle 5 (21 or 28 Day Cycle): Predose and at multiple timepoints, depending on study part.
  Cmax of LY2835219, letrozole, anastrozole, tamoxifen, exemestane, everolimus, trastuzumab, LY3023414, fulvestrant, and pertuzumab.
Number of Participants with a Complete or Partial Tumor Response (Overall Response Rate) | Baseline to study completion (estimated as 12 months)
  Number of participants with a complete or partial tumor response (overall response rate).
Progression Free Survival (PFS) | First dose to progressive disease or death of any cause (estimated as 12 months)
  Progression free survival
Change in MD Anderson Symptom Inventory (MDASI) Score from Baseline | Baseline, through study completion (estimated as 12 months)
  Change in MD Anderson (MDASI) score from baseline.
Pharmacokinetics: Area under the Curve (AUC) of LY2835219, Letrozole, Anastrozole, Tamoxifen, Exemestane, Everolimus, Trastuzumab, LY3023414, Fulvestrant, and Pertuzumab | Cycle 1 up to Cycle 5 (21 or 28 Day Cycle): Predose and at multiple timepoints, depending on study part.
  Pharmacokinetics: AUC of LY2835219, letrozole, anastrozole, tamoxifen, exemestane, everolimus, trastuzumab, LY3023414, fulvestrant, and pertuzumab.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (13):
  - Highlands Oncology Group - Duplicate 2, Rogers, Arkansas
  - University of California - San Diego, La Jolla, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University College of Phys & Surgeons, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Providence Cancer Center Oncology Hematology Care, Portland, Oregon
  - Univ of Pittsburgh Cancer Inst. (UPCI), Pittsburgh, Pennsylvania
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

REFERENCES:
- [Derived] Tolaney SM, Beeram M, Beck JT, Conlin A, Dees EC, Puhalla SL, Rexer BN, Burris HA, Jhaveri K, Helsten T, Becerra C, Kalinsky K, Moore KN, Manuel AM, Lithio A, Price GL, Chapman SC, Litchfield LM, Goetz MP. Abemaciclib in Combination With Endocrine Therapy for Patients With Hormone Receptor-Positive, HER2-Negative Metastatic Breast Cancer: A Phase 1b Study. Front Oncol. 2022 Feb 10;11:810023. doi: 10.3389/fonc.2021.810023. eCollection 2021. PMID 35223458
- [Derived] Gelbert LM, Cai S, Lin X, Sanchez-Martinez C, Del Prado M, Lallena MJ, Torres R, Ajamie RT, Wishart GN, Flack RS, Neubauer BL, Young J, Chan EM, Iversen P, Cronier D, Kreklau E, de Dios A. Preclinical characterization of the CDK4/6 inhibitor LY2835219: in-vivo cell cycle-dependent/independent anti-tumor activities alone/in combination with gemcitabine. Invest New Drugs. 2014 Oct;32(5):825-37. doi: 10.1007/s10637-014-0120-7. Epub 2014 Jun 13. PMID 24919854
- See also: Click here for more information about this study: A Study of Abemaciclib (LY2835219) in Combination With Other Therapies in Participants With Breast Cancer That Has Spread — https://www.lillytrialguide.com/en-US/studies/breast-cancer/JPBH#?postal=